CLINICAL TRIAL: NCT05854589
Title: Effect of Topical Application of Hypertonic Saline on Melanoma on Its Sizes and Number.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rafik Batroussy (Other)
Responsible Party: Sponsor-Investigator, Rafik Batroussy, Registered Pharmacist, Director, Batroussy, Rafik
Organization: Batroussy, Rafik (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 003
Record Dates: First submitted 2023-04-23; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Melanoma (Skin)
MeSH Terms: conditions — Melanoma | interventions — Water

STUDY DESIGN:
Intervention Model Description: A pilot randomized controlled study, whereas a number of patients with clinically-diagnosed skin Melanoma (any location and any stage), and who were poorly responsive to at least one cycle of conventional and standard therapy, are equally divided into 2 groups, Active and Control groups. Each patient of the Active group will have their Melanoma covered by 2 drops of water, followed by applying Sodium Chloride granules to saturate the melanoma surface then add 2 more drops of water, then cover the NaCl-granules-covered Melanoma with a bandage. The bandage will stay in place for 12 hours daily and the procedure will be repeated daily for a total of 7 consecutive days, in addition to their standard treatments they receive from their health care providers, if any. Each patient of the Control group will undergo the same treatment as the Active group patients minus the Sodium Chloride granules.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Group - Sodium Chloride Crystal Topical (Active Comparator): Each patient of the Active group will have their Melanoma covered by 2 drops of water, followed by applying Sodium Chloride granules to saturate the melanoma surface then add 2 more drops of water, then cover the NaCl-granules-covered Melanoma with a bandage. The bandage will stay in place for 12 hours daily and the procedure will be repeated daily for a total of 7 consecutive days, in addition to their standard treatments they receive from their health care providers, if any.
  Interventions: Drug: Sodium Chloride Granules
- Control Group - Plain Water topical application (Placebo Comparator): Each patient of the Control group will have their Melanoma covered by 4 drops of water, then covered by a bandage. The bandage will stay in place for 12 hours daily and the procedure will be repeated daily for a total of 7 consecutive days, in addition to their standard treatments they receive from their health care providers, if any.
  Interventions: Other: Water

INTERVENTIONS:
Drug: Sodium Chloride Granules — Sodium Chloride crystals
  Arms: Active Group - Sodium Chloride Crystal Topical
Other: Water — Plain distilled water
  Arms: Control Group - Plain Water topical application

SUMMARY:
This study evaluates the effectiveness of applying Hypertonic Saline solution directly on the Melanomas in reducing their sizes and/or number.

DETAILED DESCRIPTION:
Many previous studies have shown that Cancer cells are over-hydrated, and that Hyponatraemia exists in many cases of Cancer. The Cancer cell's viability depends on Angiogenesis and formation of blood vessels that carry water and nutrients to the rapidly-dividing Cancer cells. This study tests the hypothesis that reducing the water content of Melanoma could lead to increasing its tonicity and hence inhibiting its growth. This reduction of water content can be achieved using Osmotic Pressure differential via applying highly saline solution - made by Sodium Chloride crystals wet with water - directly on the Melanoma for a certain amount of time, thus leading to water withdrawal from Melanoma cells. While the surrounding healthy skin cells can sustain temporary dehydration, Melanoma cells could be negatively affected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically-confirmed Melanoma (any location and any stage) who have poorly responded to at least one cycle of conventional and standard therapy (Chemotherapy, Radiation or Drug therapy).
* Age 5 to 80 years old
* Life expectancy of at least 1 year
* Can understand and read English
* Lives in USA.

Patient who do not meet the Inclusion Criteria but still wish to participate will be accepted as Observational participants, but their Melanoma measurements will be not be taken into account when analyzing the Study statistically.

Exclusion Criteria:

* Skin eczema and/or other skin conditions contraindicated to skin dehydration.
* Ulcers or open wounds close to Melanoma
* Any medical condition that might cause the patient to lose consciousness
* Participants who are not residents of USA.

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Melanoma size | 6 month
  Change in Melanoma's parameters such as length and width.
Melanoma number | 6 month
  Change in Melanoma number

CONTACTS AND LOCATIONS:
Overall Officials: Rafik Batroussy, BPharm, Study Chair — Independent Researcher

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McIntyre GI. Cell hydration as the primary factor in carcinogenesis: A unifying concept. Med Hypotheses. 2006;66(3):518-26. doi: 10.1016/j.mehy.2005.09.022. Epub 2005 Nov 3. PMID 16271440
- [Background] Machado M, Salgado TM, Hadgraft J, Lane ME. The relationship between transepidermal water loss and skin permeability. Int J Pharm. 2010 Jan 15;384(1-2):73-7. doi: 10.1016/j.ijpharm.2009.09.044. Epub 2009 Sep 30. PMID 19799976
- See also: Synthetic ion transporters can induce apoptosis by facilitating chloride anion transport into cells. — https://www.nature.com/articles/nchem.2021
- See also: High Salt Inhibits Tumor Growth by Enhancing Anti-tumor Immunity. — https://www.frontiersin.org/articles/10.3389/fimmu.2019.01141/full
- See also: The osmotic passage of water and gases through the human skin. — http://royalsocietypublishing.org/doi/abs/10.1098/rspb.1932.0065
- See also: Cell swelling, softening and invasion in a three-dimensional breast cancer model. — https://www.nature.com/articles/s41567-019-0680-8
- See also: Cell Stiffness May Indicate Likelihood of Cancer Metastasis. — https://www.genengnews.com/news/cell-stiffness-may-indicate-likelihood-of-cancer-metastasis/
- See also: The Dysfunction of Metabolic Controlling of Cell Hydration Precedes Warburg Phenomenon in Carcinogenesis — https://www.longdom.org/open-access/the-dysfunction-of-metabolic-controlling-of-cell-hydration-precedes-warburg-phenomenon-in-carcinogenesis-jbb.10000e59.pdf